CLINICAL TRIAL: NCT06599177
Title: Patients with COPD: Assessment of Psychosocial Status and the Impact of Psychosocial Interventions
Brief Title: The Impact of Psychosocial Interventions in Patients with COPD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Crete (Other)
Responsible Party: Principal Investigator, Antonia Aravantinou Karlatou, Principal Investigator, University of Crete
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 56/28.03.2024
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Social Support; Intervention
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Participants will complete a questionnaire for this study and subsequently will get interviewed. Then, half of them will be randomly assigned to intervention group and control group, the intervention group participants will receive an informational leaflet that will provide information regarding psychosocial support. After, six (6) months all participants will be contacted by the P.I. to re-complete each questionnaire and repeat the interview.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): These participants will receive the informational leaflet
  Interventions: Other: Informational leaflet
- Control group (No Intervention): These participants will not receive the informational leaflet

INTERVENTIONS:
Other: Informational leaflet — An informational leaflet describing:
  * Information on benefits to which they are entitled and how to receive them.
  * Information and linkage to support services in the community.
  * Information on how to obtain health care materials (insured, uninsured).
  * Information on relevant support associations/voluntary groups in the community.
  * Information on employment programs.
  * Activation of patient's supportive social network/or referral to home help programs if they are a lonely person or in need of support.
  * Individualized assessment of the patient's needs.
  * Design of a plan for individualised psychosocial intervention (focus personal intervention).
  * Patient education about existing social support networks in the community and how to find them.
  * Educate patients about available resources in the community (benefits, services).
  * Patient referral/advocacy to community services.
  Arms: Intervention group

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is one of the most common exacerbating, non-communicable diseases. It is the third leading cause of death worldwide, causing 3.23 million deaths in 2019. Given the above, there is an international need to develop appropriate strategies for its management. COPD affects both the physical and psychosocial well-being of patients. Studies have shown that anxiety, depression, lack of social support and poor financial status are associated with more frequent exacerbations, hospital readmissions, nonadherence to treatment and worse quality of life for patients. Therefore, socioeconomic and psychological factors play a critical role in COPD. The psychosocial support of patients with COPD it is likely to be an important method for improving their health status and therefore their quality of life. The aim of this PhD thesis is to assess the psychosocial status and the impact of psychosocial information-interventions in patients with COPD. For this purpose, a prospective study of mixed methodology design (questionnaires, interviews) as well as psychosocial interventions will be conducted in patients with COPD who are attended by Pulmonary Departments of Hospitals (Outpatient Clinics, Clinics), by Local Health Units (TOMY), Regional Clinics in the prefecture of Heraklion. Interventions will include counseling for 6 months/information about services, patient benefits, support, and patients will receive a relevant form. For the implementation of the study, they will use the investigative tools (questionnaires) for the patient's health status/quality of life (SF-12-CCQ), treatment adherence (TAI), mental status (PHQ-4 includes PHQ-2 for depression and GAD-2 for anxiety) and socioeconomic status (MSPSS, FAS). Then a qualitative part will take place with an interview. At the end of 6 months the participants will be asked to answer again the same questionnaires and a partially modified interview, so that the effectiveness of the psychosocial interventions they received. Their responses will be recorded and the results will be analyzed. This study is expected to contribute to a better management of patients with COPD.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is one of the most common exacerbating, non-communicable diseases. It is the third leading cause of death worldwide, causing 3.23 million deaths in 2019. Given the above, there is an international need to develop appropriate strategies for its management. COPD affects both the physical and psychosocial well-being of patients. Studies have shown that anxiety, depression, lack of social support and poor financial status are associated with more frequent exacerbations, hospital readmissions, nonadherence to treatment and worse quality of life for patients. Therefore, socioeconomic and psychological factors play a critical role in COPD. The psychosocial support of patients with COPD it is likely to be an important method for improving their health status and therefore their quality of life. The aim of this PhD thesis is to assess the psychosocial status and the impact of psychosocial information-interventions in patients with COPD. For this purpose, a prospective study of mixed methodology design (questionnaires, interviews) as well as psychosocial interventions will be conducted in patients with COPD who are attended by Pulmonary Departments of Hospitals (Outpatient Clinics, Clinics), by Local Health Units (TOMY), Regional Clinics in the prefecture of Heraklion. Interventions will include counseling for 6 months/information about services, patient benefits, support, and patients will receive a relevant form. For the implementation of the study, they will use the investigative tools (questionnaires) for the patient's health status/quality of life (SF-12-CCQ), treatment adherence (TAI), mental status (PHQ-4 includes PHQ-2 for depression and GAD-2 for anxiety) and socioeconomic status (MSPSS, FAS). Then a qualitative part will take place with an interview. At the end of 6 months the participants will be asked to answer again the same questionnaires and a partially modified interview, so that the effectiveness of the psychosocial interventions they received. Their responses will be recorded and the results will be analyzed. This study is expected to contribute to a better management of patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a confirmed diagnosis of COPD.
* Participants should be attended by the above healthcare departments in the Heraklion Prefecture.
* Know the Greek dialect.
* Have the ability to sign a consent form.

Exclusion Criteria:

* Patients with severe and/or mental disorders.
* Patients with severe mental disability or advanced neurodegenerative disease. - Patients who do not wish to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-09-08 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Multidimensional Scale of Perceinved Social Support (MSPSS) | Through study completion, an average of a year and a half (1.5 years).
  To assess patients perceived social support, the Multidimensional Scale of Perceived Social Support (MSPSS) (Zimet et al., 1988), translated and weighted in Greek (Theofilou, 2015), will be used.The MSPSS includes 12 questions in 3 domains of perceived social support (family, friends, significant others) with 4 items in each subscale, ranging from 1-7 (likert-type) with a total score of minimum 12 and maximum 84. Higher scores indicate greater social support. Scores 12-35 indicate low perceived social support, scores 36-60 indicate moderate perceived social support, and scores 61-84 indicate high perceived social support.
Patient Health Questionnaire (PHQ-4) | Through study completion, an average of a year and a half (1.5 years).
  To assess the mental state of the patients (anxiety and depression), the Patient Health Questionnaire (PHQ-4) (Löwe et al., 2010), translated and weighted in Greek (Christodoulaki et al., 2022), will be used. The PHQ-4 is a brief assessment of anxiety and depression including 4 questions. Questions 1 and 2 are subscales of the anxiety assessment of the GAD-2 exploratory instrument, while questions 3 and. 4 are subscales of the depression assessment of the PHQ-2 exploratory instrument. The PHQ-4 includes 4 questions in the range 0-3 (likert-type) with a total score of 0 to 12. The higher the score the less anxiety/depression. A score above 3 on either indicates that further assessment with the PHQ-9 Patient Health Questionnaire or the GAD-7 Generalized Anxiety Disorder Scale should be done.
Financial Ability Scale (FAS) | Through study completion, an average of a year and a half (1.5 years).
  The Financial Ability Scale (FAS) questionnaire, translated into Greek (Koutsimpou et al., 2020), will be used to assess the financial status of the patients. The FAS includes 12 likert-type questions (ranging from no, little, moderate, good, very good).
Test of the Adherence to Inhalers (TAI) | Through study completion, an average of a year and a half (1.5 years).
  To assess patients adherence to treatment, the Test of the Adherence to Inhalers (TAI) questionnaire (Plaza et al., 2016), translated and weighted in Greek (Ierodiakonou et al., 2020), will be used.The TAI includes 12 questions ranging from 1-5 (likert type) with a total score of minimum 10 and maximum 50, which classifies patients adherence to treatment and indicates specific behavioural patterns (voluntary, involuntary, etc.) of adherence.
Sort Form (SF-12) | Through study completion, an average of a year and a half (1.5 years).
  The Sort Form (SF-12) questionnaire (Ware and Sherbourne, 1992), often used as a quality of life assessment questionnaire, translated and weighted in Greek (Kontodimopoulos et al., 2007), will be used to assess the patients health overview.The SF-12 is a short form of the SF-36 questionnaire and studies 4 domains of the patients health: physical role, physical functioning, emotional role, mental health. Each dimension is rated on a scale from 0 to 100, with 0 points representing worse health-related quality of life, and 100 points representing better health-related quality of life.
Clinical COPD Questionnaire (CCQ) | Through study completion, an average of a year and a half (1.5 years).
  For the assessment of the patients quality of life, the Clinical COPD Questionnaire (CCQ) (van der Molen et al., 2003), translated and weighted in Greek (Tsiligianni et al., 2012), (Papadopoulos et al., 2011), will be used. The CCQ includes 10 questions ranging from 0-6 (likert-type), where patients are asked to recall their experiences in the last 24 hours. The higher the score, the worse the patients health status.

CONTACTS AND LOCATIONS:
Overall Officials: Ioanna Tsiligianni, Associate professor, Study Chair — Department of Social Medicine, School of Medicine, University of Crete; Sophia Schiza, Professor of Pulmonology, Study Director — Sleep Disorders Center, Department of Respiratory Medicine, School of Medicine, University of Crete; Evangelos Karademas, Professor of Psychology, Study Director — Department of Psychology, University of Crete; Antonia Aravantinou Karlatou, Social Worker MSc, PhDc, Principal Investigator — Department of Social Medicine, School of Medicine, University of Crete
Locations (1):
- University of Crete, Heraklion, Crete, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brien SB, Stuart B, Dickens AP, Kendrick T, Jordan RE, Adab P, Thomas M. Independent determinants of disease-related quality of life in COPD - scope for nonpharmacologic interventions? Int J Chron Obstruct Pulmon Dis. 2018 Jan 9;13:247-256. doi: 10.2147/COPD.S152955. eCollection 2018. PMID 29386893
- [Background] Burney P, Jithoo A, Kato B, Janson C, Mannino D, Nizankowska-Mogilnicka E, Studnicka M, Tan W, Bateman E, Kocabas A, Vollmer WM, Gislason T, Marks G, Koul PA, Harrabi I, Gnatiuc L, Buist S; Burden of Obstructive Lung Disease (BOLD) Study. Chronic obstructive pulmonary disease mortality and prevalence: the associations with smoking and poverty--a BOLD analysis. Thorax. 2014 May;69(5):465-73. doi: 10.1136/thoraxjnl-2013-204460. Epub 2013 Dec 18. PMID 24353008
- [Background] Christodoulaki A, Baralou V, Konstantakopoulos G, Touloumi G. Validation of the Patient Health Questionnaire-4 (PHQ-4) to screen for depression and anxiety in the Greek general population. J Psychosom Res. 2022 Sep;160:110970. doi: 10.1016/j.jpsychores.2022.110970. Epub 2022 Jun 16. PMID 35728338
- [Background] Coventry PA, Gemmell I, Todd CJ. Psychosocial risk factors for hospital readmission in COPD patients on early discharge services: a cohort study. BMC Pulm Med. 2011 Nov 4;11:49. doi: 10.1186/1471-2466-11-49. PMID 22054636
- [Background] Ierodiakonou D, Sifaki-Pistolla D, Kampouraki M, Poulorinakis I, Papadokostakis P, Gialamas I, Athanasiou P, Bempi V, Lampraki I, Tsiligianni I; Greek UNLOCK group. Adherence to inhalers and comorbidities in COPD patients. A cross-sectional primary care study from Greece. BMC Pulm Med. 2020 Sep 25;20(1):253. doi: 10.1186/s12890-020-01296-3. PMID 32977779
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Kontodimopoulos N, Pappa E, Niakas D, Tountas Y. Validity of SF-12 summary scores in a Greek general population. Health Qual Life Outcomes. 2007 Sep 28;5:55. doi: 10.1186/1477-7525-5-55. PMID 17900374